CLINICAL TRIAL: NCT05808582
Title: Multicenter, Single-arm, Open Clinical Study of Chidamide in Combination With Fulvestrant in HR+/HER2-advanced Breast Cancer That Has Failed Prior CDK4/6 Inhibitor Combined With Aromatase Inhibitor Therapy
Brief Title: Chidamide Combined With Fulvestrant for HR+/HER2-advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-C37
Record Dates: First submitted 2023-03-06; First posted 2023-04-11 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Hormone Receptor-positive Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chidamide combined with fulvestrant (Experimental): fulvestrant
  Interventions: Drug: chidamide，fulvestrant

INTERVENTIONS:
Drug: chidamide，fulvestrant — chidamide combined with fulvestrant
  Other Names: Regular Visits

SUMMARY:
evaluate the efficacy and safety of chidamide combined with fulvestrant for HR+ABC

DETAILED DESCRIPTION:
This trial is a single-arm study. Designed to evaluate the efficacy and safety of chidamide combined with fulvestrant for HR+/HER2- advanced breast cancer that has failed previous CDK4/6 inhibitor combined with aromatase inhibitor therapy

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, female.
2. Both postmenopausal and premenopausal for hormone receptor positive patients, but premenopausal patients need to be given concomitant ovarian function suppression (OFS) therapy (criteria for menopause: "Judgment Criteria for Menopause after Adjuvant Therapy and Consensus on Clinical Application of Aromatase Inhibitors for Premenopausal Female Breast Cancer Patients in China").
3. Patients with HR-positive (ER-positive, PR-positive or negative) and HER2-negative breast cancer confirmed by histopathology, defined as follows.
4. Pre-enrollment disease status of non-surgically resectable locally advanced or metastatic breast cancer.
5. At least one extracranial measurable lesion as defined by RECIST V1.1 criteria or bone metastases alone.
6. Progress after previous treatment with CDK4/6 inhibitor combined with any aromatase inhibitor (after previous treatment with CDK4/6 inhibitor combined with aromatase inhibitor, you can enter the study directly or re-enter the group after chemotherapy); ; The total number of previous rescue treatments is ≤3; Previously received rescue chemotherapy ≤1 line; Time interval from the last treatment: (a) If the last treatment is endocrine therapy, it needs ≥2 weeks; (b) If the last treatment is chemotherapy, it needs ≥4 weeks;
7. ECOG PS score: 0-1.
8. Organ function meets the requirement.
9. expected survival ≥ 3 months.
10. Subjects of childbearing potential need to have a negative pregnancy test within 7 days prior to initiation of treatment and must use an appropriate method of contraception during treatment and for three months after completion of treatment.
11. Patients are fully informed and voluntarily sign an informed consent form.

Exclusion Criteria:

1. Prior treatment with any HDAC inhibitor or fulvestrant.
2. known hypersensitivity to the drug components of this trial.
3. have inflammatory breast cancer at the time of screening
4. clinical evidence or history of central nervous system metastases (CS) and/or carcinomatous meningitis, soft meningeal disease
5. inability or unwillingness to swallow medications or receive intramuscular injections
6. have gastrointestinal insufficiency or gastrointestinal disease that can significantly interfere with the absorption of study drug (e.g., uncontrolled ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
7. History of immunodeficiency, including testing positive for HIV, or having other acquired or congenital immunodeficiency disorders, or a history of organ transplantation.
8. other malignancies (except cured basal cell carcinoma of the skin, cervical carcinoma in situ and thyroid cancer) within the previous 5 years or concurrently
9. having undergone a major surgical operation or significant trauma within 4 weeks prior to initiation of treatment, or where the patient is expected to undergo major surgical treatment
10. Inability to understand or follow study guidelines and requirements.
11. Those who are judged by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from the date of informed consent to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  The overall response rate is defined as the percentage of patients with a best overall response of CR or PR relative to the appropriate analysis set
clinical benefit rate（CBR） | 2 years
  Defined as the percentage of patients who achieved complete remission (CR), partial remission (PR) and stable disease (SD) for ≥24 weeks as a percentage of the total number of patients in the analysis set.
The Number of Participants Who Experienced Adverse Events (AE) | 2 years
  Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events).

IPD SHARING:
Plan to Share IPD: No